CLINICAL TRIAL: NCT02466737
Title: Comparison of Axillary Sentinel Lymph Node Biopsy Versus no Axillary Surgery in Patients With Early-stage Invasive Breast Cancer and Breast-conserving Surgery: a Randomized Prospective Surgical Trial. Intergroup-Sentinel-Mamma (INSEMA)-Trial
Brief Title: Comparison of Axillary Sentinel Lymph Node Biopsy Versus no Axillary Surgery
Acronym: INSEMA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rostock (Other)
Collaborators: German Cancer Aid (Other); GBG Forschungs GmbH (Other)
Responsible Party: Principal Investigator, Toralf Reimer, MD PhD, Prof. Dr. Toralf Reimer, University of Rostock
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: GBG 75 / ABCSG 43
Record Dates: First submitted 2015-06-04; First posted 2015-06-09 (Estimated); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
Keywords: axillary surgery; sentinel lymph node biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- no axillary surgery (Experimental)
  Interventions: Procedure: no axillary surgery versus SLNB
- sentinel lymph node biopsy (Active Comparator): standard arm in first randomization
  Interventions: Procedure: no axillary surgery versus SLNB
- sentinel lymph node biopsy alone (Experimental)
  Interventions: Procedure: SLNB versus completion ALND
- completion axillary lymph node dissection (Active Comparator): standard arm in second randomization
  Interventions: Procedure: SLNB versus completion ALND

INTERVENTIONS:
Procedure: no axillary surgery versus SLNB — in cases with newly diagnosed breast cancer and clinically negative axillary status
  Arms: no axillary surgery; sentinel lymph node biopsy
Procedure: SLNB versus completion ALND — in cases with 1-3 macrometastases in sentinel lymph nodes
  Arms: completion axillary lymph node dissection; sentinel lymph node biopsy alone

SUMMARY:
Although there is no doubt that the presence of lymph node metastases worsens prognosis of a patient, unambiguous evidence to support lymph node dissection is still lacking. For many solid tumors, the role of lymph node dissection is yet controversial, and may depend on the tumor type and the stage of patient presentation for diagnosis. Axillary surgery for breast cancer is now considered as staging procedure that does not seem to influence breast cancer mortality. Women with breast cancer have benefitted greatly from a series of carefully performed randomized controlled trial focusing on axillary surgery. The objective of INSEMA is to show that less axillary surgery is better, in that oncological outcomes are the same and less surgical intervention will result in fewer surgical complications.

DETAILED DESCRIPTION:
Currently, axillary surgery for breast cancer is considered as staging procedure that does not seem to influence breast cancer mortality, since the risk of developing metastasis depends mainly on the biological behaviour of the primary (seed-and-soil model). Based on this, the postsurgical therapy should be considered on the basis of biologic tumor characteristics rather than nodal involvement.

The goal of the present study is to show that early-stage breast cancer patients with reduced extent of axillary surgery are not inferior regarding disease-free survival outcome compared with the standard arm. All patients will be first randomized to either no axillary surgical intervention or axillary sentinel lymph node biopsy (SLNB). Patients with SLNB and pN+(sn) status will be secondly randomized to either SLNB alone or completion axillary lymph node dissection (ALND) in cases with less than four involved nodes (1-3 macrometastases). Patients with four or more metastatic sentinel lymph nodes should undergo completion ALND.

Postoperative systemic treatment should be based on local multidisciplinary tumor board recommendation according to the current German AGO and S3 guidelines. For women who are treated with breast-conserving surgery, the most common site of local recurrence is the conserved ipsilateral breast itself. Thus, whole-breast radiation therapy after breast-conserving surgery is mandatory and should be performed according to the current guidelines (S3, AGO, DEGRO).

During follow-up, patients will be assessed for disease recurrence according to standard clinical practice. History and physical examination will be performed every 6 months for the first 36 months and yearly thereafter. Annual mammography and sonography will be required; other testing will be based on symptoms and investigator preference. The total number of patients to be randomized into the trial will be approximately 7,095. An event-driven final efficacy analysis will be performed per-protocol for two primary objectives.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to beginning breast-conserving surgery, including expected cooperation of the patients for follow-up, must be obtained and documented according to the local regulatory requirements
* Histologically confirmed unilateral primary invasive carcinoma of the breast (core biopsy or open biopsy). Multifocal or multicentric tumors are allowed if breast-conserving surgery is planned
* Age at diagnosis at least 18 years
* Preoperative imaging techniques with estimated tumor size of <5 cm (iT1/iT2 irrespective of hormone sensitivity or HER2 status)
* Clinically and sonographically tumor-free axilla prior to core biopsy (cN0/iN0)
* In cases with cN0 and iN+, a negative core biopsy or fine needle aspiration (FNA) biopsy of the sonographically suspected lymph node is required before randomization
* No clinical evidence for distant metastasis (M0)
* Planned breast-conserving surgery (R0 resection) with postoperative external whole-breast irradiation (conventional fractionation or hypofractionation)

Exclusion Criteria:

* History of malignancy within last 5 years, except curatively treated basalioma of the skin and carcinoma in situ of the cervix
* Time since core biopsy >3 months (optimal <1 month)
* Previous and already (neoadjuvant) treated invasive breast carcinoma
* Histologically non-invasive breast carcinoma
* cT3/T4 or iT3/T4 tumors
* pregnant or lactating patients
* Planned total mastectomy (e.g. multicentric tumors )
* Planned intraoperative radiotherapy (e.g. Intrabeam) or postoperative partial breast irradiation (e.g. multicatheter technique) alone; both procedures are allowed as boost techniques
* Male patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5505 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
invasive disease-free survival (IDFS) after breast-conserving surgery | 5 years
  non-inferiority question

CONTACTS AND LOCATIONS:
Overall Officials: Toralf Reimer, MD, PhD, Study Chair — University Medicine Rostock
Locations (150):
- Austria (8):
  - BGZ Dornbirn, Gynäkologie, Dornbirn
  - LKH Uni-Klinikum Graz, Gynäkologie, Graz
  - Ordensklinikum-BHS, Linz
  - Kepler Universitätsklinikum, Linz
  - KH der Barmherzigen Brüder, Saint Veit/Glan
  - Universitätsfrauenklinik Salzburg, Salzburg
  - Hanusch-Krankenhaus, Brustzentrum, Vienna
  - Landes-Krankenhaus Wolfsberg, Chirurgie, Wolfsberg
- Germany (142):
  - Ostalb-Klinikum, Brustzentrum Aalen, Aalen, Baden-Wurttemberg
  - Caritas-Krankenhaus Brustzentrum Tauberfranken, Bad Mergentheim, Baden-Wurttemberg
  - Klinikum Mittelbach Brustzentrum, Baden-Baden, Baden-Wurttemberg
  - Sana-Klinikum Biberach, Biberach, Baden-Wurttemberg
  - Krankenhaus Bietigheim, Bietigheim, Baden-Wurttemberg
  - Klinikum Böblingen, Böblingen, Baden-Wurttemberg
  - Fürst-Stirum-Klinik, Bruchsal, Baden-Wurttemberg
  - Brustzentrum Donau-Riß, Ehingen, Baden-Wurttemberg
  - Klinikum Esslingen, Esslingen am Neckar, Baden-Wurttemberg
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Frauenklinik Freudenstadt, Freudenstadt, Baden-Wurttemberg
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Städtisches Klinikum Karlsruhe, Karlsruhe, Baden-Wurttemberg
  - ViDia Christliche Kliniken, Diakonissenkrankenhaus Karlsruhe, Karlsruhe, Baden-Wurttemberg
  - St. Elisabethen Krankenhaus, Loerrach, Baden-Wurttemberg
  - Klinikum Ludwigsburg, Ludwigsburg, Baden-Wurttemberg
  - Helios Klinik Pforzheim, Pforzheim, Baden-Wurttemberg
  - Siloah St. Trudpert Klinikum, Pforzheim, Baden-Wurttemberg
  - Klinikum am Steinenberg, Reutlingen, Baden-Wurttemberg
  - Helios Klinik Rottweil, Rottweil, Baden-Wurttemberg
  - Rems-Murr Klinik, Schorndorf, Baden-Wurttemberg
  - Klinikum Tuttlingen, Tuttlingen, Baden-Wurttemberg
  - Universitätsfrauenklinik, Tübingen, Baden-Wurttemberg
  - Universitätsfrauenklinik Ulm, Ulm, Baden-Wurttemberg
  - Schwarzwald-Baar Klinikum, Villingen-Schwenningen, Baden-Wurttemberg
  - Rems-Murr Kliniken, Winnenden, Baden-Wurttemberg
  - Klinikum St. Marien, Amberg, Bavaria
  - AN regiomed Klinikum Ansbach, Ansbach, Bavaria
  - Klinikum Aschaffenburg, Aschaffenburg, Bavaria
  - Hämatologisch-onkologische Praxis, Augsburg, Bavaria
  - Klinikum Bayreuth GmbH, Frauenklinik, Bayreuth, Bavaria
  - Kreisklinik Ebersberg, Ebersberg, Bavaria
  - Gynäkologische Praxis, Eggenfelden, Bavaria
  - Klinikum Fürth, Fürth, Bavaria
  - Klinikum Kempten-Oberallgäu, Kempten (Allgäu), Bavaria
  - Klinikum Landshut, Landshut, Bavaria
  - Klinikum Fichtelgebirge gGmbH, Brustzentrum, Marktredwitz, Bavaria
  - Klinikum Memmingen, Memmingen, Bavaria
  - Klinikum der Universität München, München, Bavaria
  - Klinikum Harlaching, Frauenklinik, München, Bavaria
  - Klinikum Passau, Passau, Bavaria
  - Frauenklinik der Universität Regensburg, Caritas-Krankenhaus St. Josef, Regensburg, Bavaria
  - Klinikum Starnberg, Starnberg, Bavaria
  - Klinikum Traunstein, Traunstein, Bavaria
  - Kliniken Nordoberpfalz AG, Brustzentrum Weiden, Weiden, Bavaria
  - Rotkreuzklinik Würzburg, Würzburg, Bavaria
  - Klinikum Mitte, Missio Brustzentrum, Würzburg, Bavaria
  - Städtisches Klinikum Brandenburg, Brandenburg, Brandenburg
  - Carl-Thiem-Klinikum, Cottbus, Brandenburg
  - Ev. Krankenhaus, Frauenklinik, Ludwigsfelde, Brandenburg
  - Klinikum Ernst von Bergmann, Potsdam, Brandenburg
  - St. Joseph Stift, Bremen, City state Bremen
  - DIAKO Krankenhaus Bremen, Bremen, City state Bremen
  - Universitätsklinikum Hamburg, Brustzentrum, Hamburg, Hamburg
  - Agaplesion Diakonieklinikum, Brustzentrum, Hamburg, Hamburg
  - Gynäkologische Praxisklinik Harburg, Hamburg, Hamburg
  - Albertinen-Krankenhaus, Brustzentrum, Hamburg, Hamburg
  - Agaplesion Markus Krankenhaus, Frankfurt am Main, Hesse
  - Universitätsklinikum Brustzentrum, Frankfurt am Main, Hesse
  - Klinikum Frankfurt Höchst, Frankfurt am Main, Hesse
  - Main-Kinzig-Kliniken Gelnhausen, Gelnhausen, Hesse
  - Klinikum Hanau GmbH, Hanau, Hesse
  - Kreiskrankenhaus Bergstraße gGmbH, Heppenheim an der Bergstrasse, Hesse
  - Elisabeth Krankenhaus Kassel, Kassel, Hesse
  - Klinikum Kassel, Kassel, Hesse
  - Sana Klinikum Offenbach, Offenbach, Hesse
  - St. Josefs-Hospital, Frauenklinik, Wiesbaden, Hesse
  - Asklepios Paulinenklinik, Wiesbaden, Hesse
  - Helios Dr. Horst Schmidt Klinikum, Wiesbaden, Hesse
  - AKH Celle, Brustzentrum, Celle, Lower Saxony
  - Franziskus Hospital Harderberg, Georgsmarienhütte, Lower Saxony
  - Helios Klinikum Gifhorn, Gifhorn, Lower Saxony
  - Henriettenstiftung Frauenklinik, Hanover, Lower Saxony
  - Vinzenzkrankenhaus Hannover, Hanover, Lower Saxony
  - MHH Frauenklinik, Hanover, Lower Saxony
  - St. Bernward Krankenhaus, Hildesheim, Lower Saxony
  - Bonifatius-Hospital, Brustzentrum, Lingen, Lower Saxony
  - Euregio-Klinik Brustzentrum Nordhorn, Nordhorn, Lower Saxony
  - Agaplesion Ev. Klinikum, Brustzentrum Schaumburg, Obernkirchen, Lower Saxony
  - Klinikum Osnabrück, Osnabrück, Lower Saxony
  - Diakoniekrankenhaus, Frauenklinik, Rotenburg (Wümme), Lower Saxony
  - Klinikum Wolfsburg, Frauenklinik, Wolfsburg, Lower Saxony
  - Universität Greifswald, Frauenklinik, Greifswald, Mecklenburg-Vorpommern
  - Dietrich Bonhoeffer Klinikum, Brustzentrum, Neubrandenburg, Mecklenburg-Vorpommern
  - Universitäts-Frauenklinik, Rostock, Mecklenburg-Vorpommern
  - Helios Kliniken Schwerin, Schwerin, Mecklenburg-Vorpommern
  - Augusta-Klinik, Bochum, Nordrhein
  - Universitätsfrauenklinik Bonn, Bonn, Nordrhein
  - Marienhospital Bottrop, Bottrop, Nordrhein
  - Uniklinik Köln, Cologne, Nordrhein
  - St. Elisabeth Krankenhaus, Brustzentrum, Cologne, Nordrhein
  - Frauenklinik der H.-Heine-Universität, Düsseldorf, Nordrhein
  - Universitätsklinikum Essen Frauenklinik, Essen, Nordrhein
  - Kliniken Essen-Mitte, Essen, Nordrhein
  - Klinikum Märkische Kliniken, Brustzentrum, Lüdenscheid, Nordrhein
  - Klinikum Lünen, Brustzentrum, Lünen, Nordrhein
  - St. Franziskus-Hospital, Münster, Nordrhein
  - Universitätsklinikum Münster, Münster, Nordrhein
  - Marienkrankenhaus, Schwerte, Nordrhein
  - St. Marienkrankenhaus, Frauenklinik, Siegen, Nordrhein
  - St. Josef-Hospital, BZ Rhein-Sieg, Troisdorf, Nordrhein
  - Katharinen-Hospital, Brustzentrum, Unna, Nordrhein
  - Marien-Hospital, Wesel, Nordrhein
  - Westpfalz Klinikum, Kaiserslautern, Rhineland-Palatinate
  - BZ Mittelrhein Koblenz+Mayen, Koblenz, Rhineland-Palatinate
  - Klinikum Ludwigshafen, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Diakonissen-Stiftungs-Krankenhaus Speyer, Speyer, Rhineland-Palatinate
  - Stadtkrankenhaus Worms, Worms, Rhineland-Palatinate
  - Krankenhaus St. Elisabeth und St. Barbara, Halle, Saint
  - Universität Halle/Saale, Frauenklinik, Halle, Saint
  - Klinik St. Marienstift, Magdeburg, Saint
  - Altmark-Klinikum Brustzentrum, Salzwedel, Saint
  - Johanniter-Krankenhaus, Frauenklinik, Stendal, Saint
  - Harzklinikum, Brustzentrum Harz, Wernigerode, Saint
  - Brustzentrum Nordsachsen, Borna, Saxony
  - Diakonissenkrankenhaus, Dresden, Saxony
  - Krankenhaus St. Joseph-Stift, Dresden, Saxony
  - Universität Dresden, Frauenklinik, Dresden, Saxony
  - Städtisches Klinikum, Görlitz, Saxony
  - Universitätsklinikum Leipzig, Brustzentrum, Leipzig, Saxony
  - St. Elisabeth Krankenhaus, Leipzig, Saxony
  - Klinikum Obergöltzsch Rodewisch, Rodewisch, Saxony
  - Helios Klinik, Schkeuditz, Saxony
  - Sana-Klinik, Eutin, Schleswig-Holstein
  - DIAKO Diakonissenkrankenhaus, Flensburg, Schleswig-Holstein
  - Universitätsklinikum Schleswig-Hostein, Kiel, Schleswig-Holstein
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck, Schleswig-Holstein
  - Charite Campus Mitte, Berlin, State of Berlin
  - Sana Klinikum Berlin-Lichtenberg, Berlin, State of Berlin
  - St. Gertrauden Krankenhaus, Berlin, State of Berlin
  - DRK Kliniken Köpenick, Berlin, State of Berlin
  - Park-Klinik Weißensee, Berlin, State of Berlin
  - Evang. Waldkrankenhaus Spandau, Berlin, State of Berlin
  - DRK-Kliniken Westend, Berlin, State of Berlin
  - Krankenhaus Waldfriede, Berlin, State of Berlin
  - Helios Klinikum, Klinik für Gynäkologie, Buch, State of Berlin
  - Hufeland-Klinik Bad Langensalza, Bad Langensalza, Thuringia
  - SRH Waldklinikum, Gera, Thuringia
  - Universitätsklinikum Jena, Jena, Thuringia
  - Helios Klinikum Meiningen, Brustzentrum, Meiningen, Thuringia
  - DRK Krankenhaus, Brustzentrum, Sömmerda, Thuringia
  - SRH Zentralklinikum Suhl, Suhl, Thuringia

REFERENCES:
- [Result] Reimer T, Stachs A, Nekljudova V, Loibl S, Hartmann S, Wolter K, Hildebrandt G, Gerber B. Restricted Axillary Staging in Clinically and Sonographically Node-Negative Early Invasive Breast Cancer (c/iT1-2) in the Context of Breast Conserving Therapy: First Results Following Commencement of the Intergroup-Sentinel-Mamma (INSEMA) Trial. Geburtshilfe Frauenheilkd. 2017 Feb;77(2):149-157. doi: 10.1055/s-0042-122853. PMID 28331237
- [Result] Hildebrandt G, Stachs A, Gerber B, Potenberg J, Krug D, Wolter K, Kuhn T, Zierhut D, Sedlmayer F, Kaiser J, Reitsamer R, Heil J, Nekljudova V, Bekes I, Loibl S, Reimer T. Central Review of Radiation Therapy Planning Among Patients with Breast-Conserving Surgery: Results from a Quality Assurance Process Integrated into the INSEMA Trial. Int J Radiat Oncol Biol Phys. 2020 Jul 15;107(4):683-693. doi: 10.1016/j.ijrobp.2020.04.042. Epub 2020 May 11. PMID 32437921
- [Result] Reimer T, Stachs A, Veselinovic K, Polata S, Muller T, Kuhn T, Heil J, Ataseven B, Reitsamer R, Hildebrandt G, Knauer M, Golatta M, Stefek A, Zahm DM, Thill M, Nekljudova V, Krug D, Loibl S, Gerber B; INSEMA investigators. Patient-reported outcomes for the Intergroup Sentinel Mamma study (INSEMA): A randomised trial with persistent impact of axillary surgery on arm and breast symptoms in patients with early breast cancer. EClinicalMedicine. 2022 Nov 25;55:101756. doi: 10.1016/j.eclinm.2022.101756. eCollection 2023 Jan. PMID 36457648
- [Result] Marme F, Krieghoff-Henning E, Gerber B, Schmitt M, Zahm DM, Bauerschlag D, Forstbauer H, Hildebrandt G, Ataseven B, Brodkorb T, Denkert C, Stachs A, Krug D, Heil J, Golatta M, Kuhn T, Nekljudova V, Gaiser T, Schonmehl R, Brochhausen C, Loibl S, Reimer T, Brinker TJ. Deep learning to predict breast cancer sentinel lymph node status on INSEMA histological images. Eur J Cancer. 2023 Dec;195:113390. doi: 10.1016/j.ejca.2023.113390. Epub 2023 Oct 18. PMID 37890350
- [Result] Reimer T, Stachs A, Veselinovic K, Kuhn T, Heil J, Polata S, Marme F, Muller T, Hildebrandt G, Krug D, Ataseven B, Reitsamer R, Ruth S, Denkert C, Bekes I, Zahm DM, Thill M, Golatta M, Holtschmidt J, Knauer M, Nekljudova V, Loibl S, Gerber B. Axillary Surgery in Breast Cancer - Primary Results of the INSEMA Trial. N Engl J Med. 2025 Mar 13;392(11):1051-1064. doi: 10.1056/NEJMoa2412063. Epub 2024 Dec 12. PMID 39665649
- [Derived] Reimer T, Stachs A, Veselinovic K, Kuehn T, Heil J, Polata S, Marme F, Trapp E, Hildebrandt G, Krug D, Ataseven B, Reitsamer R, Ruth S, Denkert C, Bekes I, Stahl N, Thill M, Strittmatter HJ, Mueller T, Golatta M, Zahm DM, Holtschmidt J, Knauer M, Nekljudova V, Loibl S, Gerber B. Axillary surgery in patients with sentinel node macrometastases: secondary results of the randomized INSEMA trial. NPJ Breast Cancer. 2026 Jan 27. doi: 10.1038/s41523-026-00902-7. Online ahead of print. PMID 41593108